CLINICAL TRIAL: NCT01051336
Title: Phase I Safety and Tolerability Study of the Taris Placebo System (A Novel Bladder Drug Delivery Platform)
Brief Title: Safety and Tolerability Study of the Taris Placebo System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TARIS Biomedical, Inc. (Industry)
Responsible Party: Julie Himes, M.D. / Chief Medical Officer, TARIS Biomedical
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAR-100-101
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: TARIS Placebo; Bladder; Interstitial Cystitis; Normal Healthy Volunteers
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TARIS Placebo (Experimental)
  Interventions: Device: TARIS Placebo
- Sham Procedure (Sham Comparator)
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Device: TARIS Placebo
  Arms: TARIS Placebo
Procedure: Sham Procedure
  Arms: Sham Procedure

SUMMARY:
The aim of this protocol is to evaluate the tolerability of the Taris placebo system for the development program and to provide key safety and tolerability data for the Taris platform.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers, 18 to 55 years of age
* Body weight >100 lbs and BMI (body mass index) within the range 18-30 kg/m2
* A score of less than 11 on the pelvic pain/urgency-frequency scale (PUF)

Exclusion Criteria:

* Presence of any bladder or urethra anatomical feature that, in the opinion of the investigator, might prevent the safe placement, indwelling use, or removal of the TARIS placebo system
* History of significant urogenital surgery (any type of bladder suspension, prolapse repair, incontinence procedure, or vaginal hysterectomy)
* History of kidney stone formation
* Chronic or recurring bacterial or viral infections of the urogenital system

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability and retention of the TARIS placebo system upon insertion, 14-day exposure and removal | 14 days

SECONDARY OUTCOMES:
Subject reported symptoms | 14 days
Routine and microscopic urinalysis | 14 days
Urine culture | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj M Jain, M.D., M.B.A., Principal Investigator — Dedicated Phase I (Arizona Urology)
Locations (1):
- Phoenix, Arizona, United States